CLINICAL TRIAL: NCT07248566
Title: Effects of Cognitive Sensory Motor Training Therapy on Dexterity and Upper Limb Function in Children With Cerebral Palsy
Brief Title: Cognitive Sensory Motor Training Therapy for Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/SADIAJAVED
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Cognition; Functional activity; Dexterity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The current study will be randomized controlled trial, data will be collected from Central
  Park Teaching Hospital. The study will include 32 participants equally divided into two groups and randomly allocated. Inclusion criteria for this study will be consist of diagnosis with cerebral palsy, age 6-12, ability to participate in cognitive sensory motor training therapy, stable medical condition, and informed consent from parents/guardians. Participants with severe cognitive impairments, unstable medical condition, history of spinal . The Experimental group will receive Cognitive Sensory Motor Training Therapy and Routine Physical Therapy, while the Control group will receive Routine Physical Therapy.Cognitive Sensory Motor Training Therapy (CSMT) for 35 minutes, five times a week, over 12 weeks. Data collection will be done before and after the interventions.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): participated in Cognitive Sensory Motor Training Therapy (CSMT) for 35 minutes, five times a week, over 12 weeks. Cognitive exercise therapy combines spatial and tactile tasks to improve cognitive function, focusing on perception and sensory awareness.
  Participants completed 5 tasks, customized to their recovery progress
  Interventions: Other: Cognitive Sensory Motor Training Therapy
- Group B (Active Comparator): participants received conventional occupational therapy, consisting of many purposeful kinetic activities such as skateboard-supported arm-sliding exercises on a tabletop, picking up a ball and putting it into a basket, bi-manual placing cone, shoulder curved arch, double curved arch, arm bicycling, donut on base, putty kneading, block stacking, peg board exercise, graded pinch exercise and plastic cone stacking. Therapists could offer passive, active-assistive or active training, as deemed appropriate to the patient's ability
  Interventions: Other: conventional occupational therapy

INTERVENTIONS:
Other: Cognitive Sensory Motor Training Therapy — Cognitive Sensory Motor Training Therapy (CSMT) for 35 minutes, five times a week, over 12 weeks. Cognitive exercise therapy combines spatial and tactile tasks to improve cognitive function, focusing on perception and sensory awareness.
  Participants completed 5 tasks, customized to their recovery progress.
  Arms: Group A
Other: conventional occupational therapy — Participants received conventional occupational therapy, consisting of many purposeful kinetic activities such as skateboard-supported arm-sliding exercises on a tabletop, picking up a ball and putting it into a basket, bi-manual placing cone, shoulder curved arch, double curved arch, arm bicycling, donut on base, putty kneading, block stacking, peg board exercise, graded pinch exercise and plastic cone stacking. Therapists could offer passive, active-assistive or active training, as deemed appropriate to the patient's ability
  Arms: Group B

SUMMARY:
The current study will be randomized controlled trial, data will be collected from Central Park Teaching Hospital. The study will include 32 participants equally divided into two groups and randomly allocated. Inclusion criteria for this study will be consist of diagnosis with cerebral palsy, age 6-12, ability to participate in cognitive sensory motor training therapy, stable medical condition, and informed consent from parents/guardians. Participants with severe cognitive impairments, unstable medical condition, history of spinal cord injury or deformity, diagnosis with other neurological conditions, and visual or hearing impairments will be excluded from the study.. The Experimental group will receive Cognitive Sensory Motor Training Therapy and Routine Physical Therapy, while the Control group will receive Routine Physical Therapy.Cognitive Sensory Motor Training Therapy (CSMT) for 35 minutes, five times a week, over 12 weeks. Data collection will be done before and after the interventions.Outcome measures will include the dexterity, and upper limb function.Tools used for data collection will be Action Research Arm Test and Box and Block Test. Data analysis will utilize SPSS version 25.00.

DETAILED DESCRIPTION:
Cerebral palsy defined as a neuro-impairment with motor disability caused by a non- progressive defect or lesion of the immature brain. Cerebral palsy (CP) impact approximately

1 in 500 children worldwide, affecting motor function, muscle tone, and coordination.

Children with CP will experience limitations in daily activities, social participation, and quality of life due to impaired upper limb function. To address this, rehabilitation strategies will focus on enhancing dexterity, and upper limb function. The aims of the study is to examine the effects of cognitive sensory motor training therapy on dexterity and upper limb function in children with CP. The current study will be randomized controlled trial, data will be collected from Central Park Teaching Hospital. The study will include 32 participants equally divided into two groups and randomly allocated. Inclusion criteria for this study will be consist of diagnosis with cerebral palsy, age 6-12, ability to participate in cognitive sensory motor training therapy, stable medical condition, and informed consent from parents/guardians. Participants with severe cognitive impairments, unstable medical condition, history of spinal cord injury or deformity, diagnosis with other neurological conditions, and visual or hearing impairments will be excluded from the study.. The Experimental group will receive Cognitive Sensory Motor Training Therapy and Routine Physical Therapy, while the Control group will receive Routine Physical Therapy.Cognitive Sensory Motor Training Therapy (CSMT) for 35 minutes, five times a week, over 12 weeks. Data collection will be done before and after the interventions.Outcome measures will include the dexterity, and upper limb function.Tools used for data collection will be Action Research Arm Test and Box and Block Test. Data analysis will utilize SPSS version 25.00.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years with cerebral palsy
* Diagnosis confirmed by pediatric neurologist or rehabilitation specialist
* Ability to follow simple instructions and participate in therapy sessions.
* Participants had to be able to focus attention on demonstrate level II and III on the Gross
* Motor Function Classification Scale (GMFCS)
* Level II or III on the Manual Ability Classification System (MACS)

Exclusion Criteria:

* Visual impairment or hearing defect
* Severe cognitive decline and aphasia
* Contractures that could limit the patient from maintaining the extended arm in a comfortable position,

Ages: 6 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test: | The test can be completed in an average of 10 minutes but requires specific materials
  The ARAT is a standardized measure of the upper extremity (arm and hand) function based
  on four movements
  : grasping, grip-ping, pinching and gross movements of shoulder,elbow and fingers. ARAT has an ordinal 4-point scale (0-3) for 19 items. Scoring is determined as follows: 0, patient cannot perform any part of task;1, patient is able to lift the object completely from the platform; 2, function is performed fully but clumsily or with great difficulty; and 3, the movement is performed normally. The maximum score for each arm is 57 points.
Box and Block Test: | The number moved in 60 seconds is the recorded score.
  The box and block test 13 will be used to evaluate gross manual dexterity. The setup consists of two adjacent boxes of the same size (53.7 × 25.4 × 8.5cm), one of them filled with 150 blocks (2.5 cm 3).Between the two boxes, there is a partition 15.2 cm in height. The patient must move blocks one by one from one box to the other, over the partition.

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Javed, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Asif Jvaed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi W. Effects of Cognitive Exercise Therapy on Upper Extremity Sensorimotor Function and Activities of Daily Living in Patients with Chronic Stroke: A Randomized Controlled Trial. Healthcare (Basel). 2022 Feb 24;10(3):429. doi: 10.3390/healthcare10030429. PMID 35326907